CLINICAL TRIAL: NCT02975427
Title: Abdominal Bioelectric Impedance for Follow-up of Dieters: A Prospective Study
Brief Title: Bioimpedance Analysis for Follow-up of Dieters
Acronym: BIA
Status: Completed | Type: Observational
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Yusuf Bozkuş, Dr., Baskent University Ankara Hospital
Other Study IDs: KA12/192
Record Dates: First submitted 2016-10-27; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Diet; Abdominal bioelectrical impedance analysis; Anthropometry; Insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diet group: All participants were prescribed an appropriate diet with caloric restriction and an exercise program and underwent a follow-up examination 3±1 months later.
  Interventions: Other: Diet group

INTERVENTIONS:
Other: Diet group — All participants were prescribed an appropriate diet with caloric restriction and an exercise program and underwent a follow-up examination 3±1 months later.

SUMMARY:
Prospective, single arm, dietary intervention study.

DETAILED DESCRIPTION:
This prospective study was conducted during the period from December 2011 through June 2013 in the Department of Endocrinology and Metabolism of Başkent University.

We enrolled 185 participants who were admitted to hospital for weight loss therapy. After initial evaluation, all participants were prescribed an appropriate diet with caloric restriction and an exercise program and underwent a follow-up examination 3±1 months later. At the end of the follow up, 103 participants attended to the research. Anthropometric, bioimpedance and laboratory measurements performed at baseline and second visit. We calculated the difference in anthropometric, bioimpedance and laboratory measurements between the first and second evaluations. Correlation analysis, multivariate linear regression analysis and receiver operating characteristic analysis performed to assess associations of laboratory metabolic variables with a decrease in anthropometric and bioimpedance analysis (BIA) measures, after diet and/or exercise therapy. The secondary aim was to determine whether abdominal BIA was better than simple anthropometric measurements and conventional BIA for assessing changes in metabolic variables.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 70 years without chronic disease, cancer, a pacemaker, cardiac valve replacement, malabsorption syndrome, previous history of gastrointestinal surgery, thyroid disease, pregnancy, or a history of surgery during the previous 3 months.

Exclusion Criteria:

* Participants receiving oral antidiabetic drugs, insulin, any treatment for obesity, steroids or hormonal drugs, over-the-counter drugs for weight loss, any kind of phytodrug, or any drug that could affect glucose metabolism. We also excluded patients who used any of these drugs after the initial evaluation.
* Participants who, at the second visit, reported that they failed to adhere to the diet.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred and eighty five participants who were admitted to hospital for weight loss therapy enrolled to the study. After initial evaluation, all participants were prescribed an appropriate diet with caloric restriction and an exercise program and underwent a follow-up examination 3±1 months later. A total of 134 participants reported for the second visit; 51 did not. Thirty one participants who, at the second visit, reported that they failed to adhere to the diet were excluded from the analysis . Ultimately, data from 103 participants who reported that they adhered to the diet were included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Value of abdominal BIA for the follow up of dieting individual | 3 months (plus or minus 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Bozkuş, Dr., Principal Investigator — Baskent University Ankara Hospital

IPD SHARING:
Plan to Share IPD: No